CLINICAL TRIAL: NCT01572194
Title: Predictive Value of PIIINP Urinary for the Development of Chronic Renal Failure in Patients With Cystic Fibrosis After Lung Transplantation.
Brief Title: Predictive Value of PIIINP Urinary for the Development of Chronic Renal Failure in Patients With Cystic Fibrosis After Lung Transplantation (MUCO-IRC)
Acronym: MUCO-IRC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: no more recruitment in the centers
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RC11_0215
Record Dates: First submitted 2012-03-28; First posted 2012-04-06 (Estimated); Last update posted 2018-04-23 (Actual); Status verified 2017-05

CONDITIONS: Lung Transplantation; Cystic Fibrosis; Renal Failure
Keywords: CF
MeSH Terms: conditions — Cystic Fibrosis; Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: Urinary levels of PIIINP as a marker of changes in renal function — The act under consideration is the determination of PIIINP urinary. The aim of the study is to show the predictive value of PIIINP urinary in assessing renal function in patients with mucoviscidosis receiving a lung transplant.

SUMMARY:
Chronic renal failure is a serious complication of lung transplantation especially in patients with cystic fibrosis. Their medical history prior to the Lung Transplantation has already exposed to kidney damage. Post-lung transplantation, these patients are subjected to renal toxicity anticalcineurins they receive large doses.

The measurement of renal function of patients by formula to estimate GFR in routine use is unreliable and other markers seem indispensable.

The purpose of this study is to evaluate two markers, PIIINP (Procollagen III aminoterminal peptide N), whose urinary levels was correlated to the intensity of fibrosis in different types of kidney disease.

ELIGIBILITY:
Inclusion Criteria:

* Bearer of lung transplantation (single or double lung, with or without associated cardiac transplantation)
* Suffering from cystic fibrosis
* Aged 18 and over
* With at least 6 months of transplantation
* Having a glomerular filtration rate measured by technical radionuclide > 30 ml / min
* Having given written consent to the study Patients meeting these criteria will enter in the "organic" in the study (determination of PIIINP urinary)

Exclusion Criteria:

* Lung transplantation for a condition other than cystic fibrosis
* Patient refused follow-up
* Patients with advanced liver disease (conditions that interfere with the assay of PIIINP)
* Minor
* Pregnant women,
* Major Trust, benefiting from a regime of legal protection (guardianship, trusteeship, safeguarding justice.
* Patient unable to grant informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2012-04; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
The correlation between the rate of urinary PIIINP inclusion in the study and the variation of the isotopic measurement of GFR over the 2 year study | 3 years

SECONDARY OUTCOMES:
Description of histological lesions present after transplantation from renal biopsies performed in all patients with chronic renal failure defined by a GFR between 30 and 60 ml / min and / or proteinuria> 1 g / d. | 3 years
Correlation between the rate of PIIINP urinary and the rate of first and second intensity of renal fibrosis histologically assessed renal biopsies that have been conducted in patients. | 3 years
Correlation between the rate of urinary PIIINP and glomerular filtration rate measured by scintigraphy Chrome-EDTA at study entry and after 2 years of follow-up | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Hourmant, Nantes, France